CLINICAL TRIAL: NCT05258383
Title: Personalized Estimation of Doses Delivered During Image Guided Radiation Therapy Tests
Acronym: ELISA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP210583; APHP210583 (Other: Assistance Publique-Hôpitaux de Paris)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lung Neoplasm; Pelvic Neoplasm; Breast Cancer; Cancer, Otorhinolaryngeal; Cancer Pediatric
Keywords: Image guided radiation therapy; dosimetry; X-rays
MeSH Terms: conditions — Lung Neoplasms; Pelvic Neoplasms; Breast Neoplasms; Otorhinolaryngologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Lung Neoplasm patients: Lung Neoplasm patients (adults)
  Interventions: Other: 3D maps of physical doses
- Pelvic Neoplasm patients: Pelvic Neoplasm patients (adults)
  Interventions: Other: 3D maps of physical doses
- Breast Cancer patients: Breast Cancer patients(adults)
  Interventions: Other: 3D maps of physical doses
- Ear Nose and Throat (ENT) Cancer patients: Ear Nose and Throat (ENT) Cancer patients (adults)
  Interventions: Other: 3D maps of physical doses
- Pediatric Cancer patients: Pediatric cancer patients (under 18 years-old) : neurologic cancer , abdomen cancer, Thorax cancer, Ear Nose and Throat (ENT) Cancer
  Interventions: Other: 3D maps of physical doses

INTERVENTIONS:
Other: 3D maps of physical doses — 3D maps of physical doses delivered to organs by positioning imaging will be calculated based on the patient's CT image used by the treatment planning system (dosimetric calculation performed by Monte Carlo method).

SUMMARY:
In image-guided radiotherapy (IGRT), the repeated and increasingly intensive use of on-board positioning imaging, using 2D or 3D Mega-Volt (MV) or kilo-Volt (kV) imaging devices (cone-beam or CBCT scanners), is leading the international medical community to question the potential impact of these additional doses delivered to the patient, especially in at-risk populations such as children and young adults. The doses delivered to the patient by positioning imaging are still relatively unknown, due to the lack of experimental means and software available in clinical routine to easily and accurately evaluate these doses.

The main objective is to estimate by personalized Monte Carlo calculation the physical doses delivered to the patient's organs by the onboard imaging systems during their radiotherapy treatment. The obtained imaging doses will be compared according to different irradiation scenarios commonly used in clinical routine as well as according to the treated location.

DETAILED DESCRIPTION:
The study will consist of 2 successive steps:

* Step 1 : for a set of patients selected in the clinical centers participating in the study, 3D maps of physical doses delivered to organs by positioning imaging will be calculated based on the patient's CT image used by the treatment planning system (dosimetric calculation performed by Monte Carlo method).
* Step 2/ all the new dosimetric data, average organ doses and dose volume histogram, will be the subject of a more global analysis, which will be returned to the project's clinical partner centers.

ELIGIBILITY:
Inclusion Criteria:

* IGRT (Image Guided Radiation Therapy) treatments considered: lung, pelvic (prostate), breast, ENT and pediatric cancers
* Treatment modalities: linac + daily kV-CBCT (kilo-Volt ConeBeam CBCT) and linac + weekly kV-CBCT + daily 2-Dimensional-kilo-Volt (2D-kV) (adult: lung, prostate, breast, Ear Nose and Throat (ENT); pediatric: neuro, ENT, thorax and abdomen); Cyberknife + daily 2D-kV (adult lung); Tomotherapy + daily MV-CBCT (Mega-Volt ConeBeam CBCT) (adult prostate, breast, ENT; pediatric ENT, thorax and abdomen)

Exclusion Criteria:

* Patient who has undergone a treatment discontinuation or modification (re-planning) of treatment with an impact on the IGRT protocol.
* Patient for which details on the imaging procedures used during treatment or DICOM files (DICOM CT, DICOM RTstruct) are incomplete will not be included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients (Lung Neoplasm, Breast Cancer, Cancer Ear Nose and Throat / ENT); Male patients (Lung Neoplasm, Pelvic Neoplasm, Cancer Ear Nose and Throat / ENT); Pediatric cancer patients.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2025-05-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
Global analysis of 3D mapping of physical doses delivered to organs by positioning imaging. | One year after end of data collection
  Global analysis of 3D mapping of physical doses delivered to organs by positioning imaging. These analyses will aggregate the Doses Volumes Histograms (HDV) by organs of interest as well as the mean dose to 10% (D10), 50% (D50) and 90% (D90) metrics for these same organs to form an individual dosimetric report.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GIRAUD, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (9):
- France (9):
  - Institut de Radiothérapie et Radiochirurgie H. Hartmann, Levallois-Perret, Hauts-de-Seine
  - Hôpital Henri Mondor - AP-HP, Créteil, Val-de-Marne
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - Groupe AMETHYST, Colombes
  - Institut Curie, Paris
  - Hôpital Saint-Louis - AP-HP, Paris
  - Hôpital La Pitié Salpêtrière - AP-HP, Paris
  - Hôpital européen Georges-Pompidou AP-HP, Paris
  - Hôpital Tenon - AP-HP, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).